CLINICAL TRIAL: NCT03761719
Title: The Influence of HDL Function on Cognitive Function and Brain Structures in Older People With Diabetes Mellitus
Brief Title: The Influence of HDL Function on Cognitive Function
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Timothy Kwok, Professor, Chinese University of Hong Kong
Other Study IDs: 2018.032
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Older People With Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Older people with diabetes mellitus are at risk of cognitive decline and dementia. We therefore propose to examine the potential influence of HDL function on global cognitive function and brain structures in older people with DM.

ELIGIBILITY:
Inclusion Criteria:

Participants with DM

Exclusion Criteria:

Participants refuse blood taking

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: DM patients
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Neurocognitive test domain scores | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong